CLINICAL TRIAL: NCT00320905
Title: Smart Heart Study: Cognitive Benefits of Cardiac Rehabilitation
Status: Completed | Type: Observational
Sponsor: Summa Health System (Other)
Responsible Party: Donna Waechter, Ph.D., Summa Health System
Other Study IDs: RP#05094
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Cardiovascular Disease
Keywords: Cardiac Rehabilitation; Cognitive functioning; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Observational — No intervention

SUMMARY:
The proposed study will be the first to examine whether changes in blood flow patterns within the brain account for the possible cognitive benefits of CR. A clearer understanding of this possibility may provide key insight into the way CVD affects the brain, help identify effective treatments, help a greater number of patients return to work, and improve quality of life.

DETAILED DESCRIPTION:
Based on recent patient referrals, we expect that 30 participants will subsequently enroll in CR and 30 will not. CR patients will complete standardized neuropsychological tests (45-60 minutes) and Transcranial Doppler (30-40 minutes) during their first and last week in the CR program. Patients who do not enroll in CR will undergo testing at similar intervals to serve as a matched control group. Standard medical records will be collected for participants in both groups to obtain demographic and medical information. CR-specific medical records will also be collected to obtain information about possible mechanisms for cognitive benefits (e.g. improved stress test performance, reduced blood pressure, etc.). All participants will be compensated for their time.

ELIGIBILITY:
Inclusion Criteria:

- 50 to 85 years of age, able to communicate in English, history of heart disease

Exclusion Criteria:

- history of significant neurological disorders, such as stroke, Alzheimer's disease, or severe head injury significant psychological problems such as schizophrenia or bipolar disorder

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2006-03; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Josephson, MD, Study Director — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States